CLINICAL TRIAL: NCT04384497
Title: Convalescent Plasma for Treatment of COVID-19: An Exploratory Dose Identifying Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Joakim Dillner (Other)
Collaborators: Danderyd Hospital (Other); Karolinska University Hospital (Other); Karolinska Institutet (Other)
Responsible Party: Sponsor-Investigator, Joakim Dillner, Professor of Infectious Disease Epidemiology; Director of R&D, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP2
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: COVID-19
Keywords: COVID-19 convalescent plasma treatment; SARS-CoV-2 infection; Dosing; Safety; Effectiveness
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Serotherapy

STUDY DESIGN:
Intervention Model Description: An open, non-randomised controlled, safety and dose identifying clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Convalescent plasma treatment (Experimental): Participants will receive 200 ml convalescent plasma daily until SARS-CoV-2 is no longer detectable in the blood up to a maximum of 7 CP infusions. CP will be given as a slow infusion over 1 hour. Patients will be monitored for adverse events, especially allergic reactions.
  Interventions: Biological: SARS-CoV-2 convalescent plasma

INTERVENTIONS:
Biological: SARS-CoV-2 convalescent plasma — Treatment with convalescent plasma (200ml, up to a maximum of 7 CP infusions). Plasma from consenting individuals who have recovered from SARS-CoV-2 infection.

SUMMARY:
Convalescent plasma has been shown to be safe and effective for treatment of several diseases. Preliminary data indicates that it is safe and effective for treatment of COVID. However, data is limited to small studies and case series on severely ill patients.

In a preliminary safety study 10 patients with severe COVID-19, defined as requiring supplementary oxygen, having fever and a duration of illness less than 11 days were treated with 200 ml of CP. CP was given as a slow infusion without obvious adverse events. Eight patients had viremia. One patient rapidly cleared the virus and recovered following CP treatment. CP infusion did not appear to clear viremia in 7/8 patients. Five of these were eventually admitted to ICU. Thus CP did not appear to cause acute toxicity but did not seem to be effective at the dose used. Viremia seemed to be a marker of a high risk of disease progression The proposed study thus aims to treat a high risk population identified by having viremia irrespective of but hopefully before they develop pulmonary injury such that they require supplementary oxygen therapy. Moreover the dose of plasma will be increased incrementally with the aim of clearing viremia as our initial study indicates that continued viremia is driving COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Admitted to a study hospital
* Active COVID-19 defined as symptoms + SARS CoV-2 identified from upper or lower airway samples
* Negative pregnancy test taken before inclusion and use of an acceptable effective method of contraception until treatment discontinuation if the participant is a woman of childbearing potential
* Written informed consent after meeting with a study physician and ability and willingness to complete follow up

Exclusion Criteria:

* No matching plasma donor (Exact matching in both the ABO system is required)
* Unavailability of plasma
* Significant growth of alternative lower airway pathogen such as Streptococcus pneumoniae or Haemophilus influenzae in sputum
* Estimated glomerular filtration rate <60 (kidney failure stage III or more)
* Pregnancy (urinary-hcg)
* Breast feeding
* History of severe allergic reactions to foods or other substances that the donor may have been exposed to (for example severe peanut allergy)
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Number and proportion of patients with progression to ventilation or sustained requirement of supplementary oxygen therapy | Measured in the first 28 days after inclusion.
  Progression to non-invasive or invasive ventilation or a sustained requirement of 15L of supplementary oxygen therapy in patients that are not eligible for intensive care treatment.

SECONDARY OUTCOMES:
Adverse events | The reporting period for AEs starts at inclusion and ends at the final follow-up visit 2 months after inclusion.
  Adverse reactions and serious adverse reactions. The safety of the intervention will be assessed with regard to AEs, baseline medical conditions, and findings from the physical examination and laboratory tests. Possible adverse events will be elicited using a modification and Swedish translation (appendix 6) of Common Terminology Criteria for Adverse Events v5.0 and they will be continuously reported to the sponsor. Adverse events related to convalescent plasma therapy shall be followed to assess reversibility.
Dose of plasma needed to clear viremia | 28 days
  Measured as doses of convalescent plasma administered (1-7 infusions, 200ml).
Clearance of viremia | 6 months.
  SARS-CoV-2 RNA detection by PCR in blood or serum. Blood samples for immunological analyses and serology will be taken daily until discharge, on day 28, and at 6 months.
Fever and symptoms | Until discharged from the hospital, up to 2 months
  Time to resolution of fever and symptoms. Breathing rate, peripheral oxygen saturation (measured with pulse oximetry after 20 minutes of rest), oxygen use, pulse, blood pressure, body temperature and mental state will be monitored 3 times/day while hospitalized.
Inflammatory parameters | Until discharged from the hospital, up to 2 months
  Time to normalization of inflammatory parameters. Blood samples for inflammatory parameters will be taken daily until normalized or discharged from the hospital.
Antibody response to SARS-CoV-2 | 6 months
  Characterization of the antibody response to SARS-CoV-2. Blood samples for immunological analyses and serology will be taken daily until discharge, on day 28, and at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Ursing, MD, PhD, Principal Investigator — Danderyd Hospital
Locations (2):
- Sweden (2):
  - Danderyd Hospital, Danderyd, Stockholm County
  - Karolinska University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
The investigators will be sharing the data, but the management plan is being designed.
Supporting Information: Study Protocol